CLINICAL TRIAL: NCT04500197
Title: A Single-centre Prospective Observational Study of MIcrocirculatory Perfusion Alterations in Severe Burn Injury
Brief Title: A Study of MIcrocirculatory Perfusion Alterations in Severe Burn Injury
Acronym: MIPA
Status: Completed | Type: Observational
Sponsor: Maasstad Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: L2015126
Record Dates: First submitted 2019-09-20; First posted 2020-08-05 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Microcirculation; Burns; Resuscitation
Keywords: microcirculation; burns; resuscitation
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective of our study is to focus on the efficiency of standard fluid resuscitation in promoting tissue perfusion in severe burns patients (>15% TBSA). The incidence of microcirculatory perfusion alterations, according to a predefined arbitrary cut off value, in patients with severe burns injury (>15%TBSA) will be assessed during standard resuscitation in the first 24 hours.

Secondary objectives are to assess differences in microcirculatory perfusion alterations between early (<12 hours post burn injury) and late standard resuscitation (>12 hours post burn injury) with addition of albumin to the regime.

And to measure several biomarkers of glycocalyx shedding, oxidative stress and inflammation.

DETAILED DESCRIPTION:
Rationale: There are valid concerns that resuscitation in burns shock is inadequate. A tendency to over resuscitate patients seem to exist. Current guidelines were developed 35 years ago and clinical burn resuscitation has not advanced significantly, despite ongoing research. The main goal of resuscitation is achieving organ perfusion and tissue oxygenation. Inadequate fluid resuscitation of severe acute burns may result in hypovolemic shock and death. Excessive fluid resuscitation may result in fluid overload, lung edema, intra-abdominal hypertension, abdominal compartment syndrome and burn depth conversion with increased requirement for escharotomies, fasciotomies and skin grafting. Monitoring of adequacy of resuscitation in burns patients has always been guided by systemic hemodynamic variables (macro circulation) like blood pressure, heart rate, stroke volume and urinary output, being urine output the major indicator of successful resuscitation. Whether these end points are successful in achieving adequate perfusion and oxygen transport to the tissues is unknown and relies on the assumption that there is a hemodynamic coherence between the macro and microcirculation whereby improving the macro circulation causes a parallel improvement in the microcirculation Objective: The main objective of our study is to focus on the efficacy of standard fluid resuscitation in promoting tissue perfusion.

Study design: Single-center, prospective, observational clinical study in the Maasstad Hospital.

Study population: All adult patients who are admitted to the Intensive Care Unit with severe burns over 15%TBSA and resuscitated with the standard resuscitation protocol will be included.

Main study parameters/endpoints: Measurement of sublingual microcirculation with vessel density and flow parameters. Also skin perfusion maps (Laser Speckle Imaging) will be recorded. Blood and urine samples will also be used for measuring glycocalyx shedding products.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

Microcirculation assessment and laser speckle imaging are non-invasive procedures, and there are negligible risks. Blood tests will be used for measuring glycocalyx shedding products, this is an invasive procedure which may increase the risk of contamination, patient discomfort and in some extreme cases blood sample collection may be a burden on patient haemoglobin levels which is prone to decrease in critical patients. Assessment is essential for determining whether action is required to change our existing resuscitation regime for critically ill burned patients. If the results show that the current resuscitation regime is suboptimal, then motivation for changing the existing practice can lead to improved clinical care and a reduction in over- or under resuscitation in the ICU environment with its potential harmful effects.

The risks associated with participation can be considered negligible and the burden can be considered minimal in this observational study. The patients taking part in this study will have no direct benefit.

ELIGIBILITY:
Inclusion Criteria:

1. ICU admission with a severe burn injuries of ≥15% TBSA
2. ≥ 18 years of age
3. Receiving standard resuscitation protocol for severe burn injury
4. Post burn time up to a maximum of 24 hours

Exclusion Criteria:

1. Informed consent not obtained
2. (suspected) generalised infection
3. Other traumatic injury, which is supposed to generate a systemic inflammatory response eg severe fractures, or other types of shock as a result of massive bleeding
4. Patients unlikely to survive >24 hours
5. Decision not to initiate treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 patients admitted to the ICU with a severe burn ≥15% TBSA will be given standard resuscitation care and will be included
Sampling Method: Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2020-09-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Measurement of microcirculatory perfusion alterations in severe burns patients during standard fluid resuscitation. | Changes in perfusion parameters will be measured on admission (time zero, T=0), four hours after admission (T=4), eight hours after admission (T=8), twelve hours after admission (T=12) and twenty-four hours after admission (T=24
  The main objective of our study is to measure standard microcirculatory perfusion parameters during standard resuscitation at different time points after a severe burn injury. These perfusion parameters are total vessel density (TVD), proportion of perfused vessels (PPV), functional capillary density (FCD) and focus depth.

SECONDARY OUTCOMES:
Microcirculatory perfusion alterations after administration of albumin. | Changes in microcirculatory perfusion parameters will be measured directly after administration of albumin. This will be 12 hours after starting fluid resuscitation.
  Secondary objectives are to measure changes in standard microcirculatory parameters before and after administration of albumin. Albumin will be administered 12 hours after admission of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Can Ince, Prof, Study Director — Erasmus Medical Center
Locations (1):
- Maasstad Hospital, Rotterdam, Zuid Nederland, Netherlands